CLINICAL TRIAL: NCT00168038
Title: An Open-label, Multicenter Study on the Efficacy and Safety of IgPro10 in Patients With Chronic Immune Thrombocytopenic Purpura (ITP)
Brief Title: Treatment of Chronic Immune Thrombocytopenic Purpura (ITP) With Intravenous Immunoglobulin IgPro10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLB03_003CR; 2004-000537-11 (EudraCT Number)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-10

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Chronic Immune Thrombocytopenic Purpura; Chronic Idiopathic Thrombocytopenic Purpura; Werlhofs Disease; Autoimmune Thrombocytopenia; Immunglobulin Intravenous; Chronic ITP; Platelet count; Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — Immunoglobulins, Intravenous

ARMS (1):
- IgPro10 (Experimental)
  Interventions: Biological: Immunoglobulin Intravenous (Human)

INTERVENTIONS:
Biological: Immunoglobulin Intravenous (Human) — A dose of 1 g IgG per kg body weight (bw) administered on two consecutive days resulting in the total treatment dosage of 2 g IgG per kg bw.
  Other Names: Privigen; IgPro10

SUMMARY:
The purpose of this study is to evaluate the efficacy, tolerability and safety of IgPro10 in the treatment of patients with chronic immune thrombocytopenic purpura (ITP). The main efficacy parameter is the proportion of patients responding to treatment by an increase of platelet count to ≥ 50 x 10^9/L.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of chronic ITP defined by: Failure to find other causes of thrombocytopenia; Platelet count ≤ 150 x 10^9/L over 6 months or response to a previous treatment with subsequent decrease in platelet count even if duration of chronic ITP is less than 6 months
* Platelet counts ≤ 20 x 10^9/L

Key Exclusion Criteria:

* Planned splenectomy throughout the study period
* Treatment with IVIG or anti-D immunoglobulin within 3 weeks prior to screening
* Treatment with immunosuppressive or other immunomodulatory drugs within 3 weeks prior to screening
* Treatment with intravenous steroids within 10 days prior to screening
* Change of oral steroid treatment within 15 days prior to screening
* Patients with known or suspected hypersensitivity to immunoglobulins or previous severe side effects to immunoglobulin therapy
* Abnormal results in the following laboratory parameters: Hemoglobin < 10 g/dL; Total bilirubin > 1.5 x upper normal limit; ALAT > 2.5 x upper normal limit; ASAT > 2.5 x upper normal limit; Creatinine > 1.5 x upper normal limit; Urea > 1.5 x upper normal limit
* Positive direct Coombs test
* Patients with one of the following concomitant diseases Clinical active SLE Known or suspected HIV infection Acute hepatitis Clinically active chronic hepatitis Lymphoproliferative disease Heart failure Grade III or IV according to the New York Heart Association classification
* Any other concomitant disease that has influence on the clotting system (i.e. hemophilia)

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-12; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Othmar Zenker, MD, Study Director — CSL Behring
Locations (17):
- Study Site, Berlin, Germany
- Study Site, Rome, Italy
- Poland (6):
  - Study Site, Bialystok
  - Study Site, Gdansk
  - Study Site, Lodz
  - Study Site, Poznan
  - Study Site, Warsaw
  - Study Site, Wroclaw
- Russia (4):
  - Study Site, Moscow
  - Study Site (19), Saint Petersburg
  - Study Site (20), Saint Petersburg
  - Study Site (21), Saint Petersburg
- Ukraine (4):
  - Study Site, Dnipropetrovsk
  - Study Site (02), Kyiv
  - Study Site (03), Kyiv
  - Study Site, Lviv
- Study Site, Taunton, United Kingdom

REFERENCES:
- [Result] Robak T, Salama A, Kovaleva L, Vyhovska Y, Davies SV, Mazzucconi MG, Zenker O, Kiessling P; International Privigen in ITP Study Group. Efficacy and safety of Privigen, a novel liquid intravenous immunoglobulin formulation, in adolescent and adult patients with chronic immune thrombocytopenic purpura. Hematology. 2009 Aug;14(4):227-36. doi: 10.1179/102453309X439773. PMID 19635187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed as a multicenter study at 17 centers, 6 in Poland, 4 in the Ukraine, 4 in Russia, 1 in Germany, 1 in Italy and 1 in the United Kingdom (UK).
Pre-assignment Details: One enrolled subject was withdrawn prior to receiving treatment due to a non-fatal adverse event. This subject was not included in the analyses.
Groups:
- IgPro10: All subjects treated with IgPro10
Period: Overall Study
Arm/Group | IgPro10
Started | 57
Completed | 55
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Therapy failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | IgPro10
Number analyzed (Participants) | 57
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 23
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 57
Weight [Mean (Standard Deviation); unit: kg] | 74.0 (15.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.69 (4.56)

OUTCOME MEASURES:

1. Primary Outcome: Platelet Response
Description: The platelet response rate is defined as the percentage of subjects responding to treatment with an increase of platelet count from ≤ 20 x 10^9/L to ≥ 50 x 10^9/L within the specified time frame.
Time Frame: 7 days
Population: Intention to treat (ITT) analysis. The ITT population comprised all subjects who received at least once study medication.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | IgPro10
Number analyzed (Participants) | 57
Percent of participants | 80.7 [69.2 to 89.3]

2. Secondary Outcome: Regression of Hemorrhage (Skin)
Description: Number of subjects with a decrease in the severity of bleeding from baseline (prior to first infusion) on at least one post-infusion assessment during the study period (e.g., a change from moderate to mild or a change from mild to none). Regression of hemorrhages was tabulated separately for the organ systems skin, oral cavity, genitourinary tract, nose, and internal.
Time Frame: up to 29 days
Population: The number of participants analyzed represents the number of subjects in the ITT population with skin bleeding at baseline and respective post-baseline assessment.
Measure: Number; unit: participants
Arm/Group | IgPro10
Number analyzed (Participants) | 36
participants | 31

3. Secondary Outcome: Regression of Hemorrhage (Oral Cavity)
Description: as for outcome 2
Time Frame: 29 days
Population: The number of participants analyzed represents the number of subjects in the ITT population with oral cavity bleeding at baseline and respective post-baseline assessment.
Measure: Number; unit: participants
Arm/Group | IgPro10
Number analyzed (Participants) | 11
participants | 11

4. Secondary Outcome: Regression of Hemorrhage (Genitourinary Tract)
Description: as for outcome 2
Time Frame: 29 days
Population: The number of participants analyzed represents the number of subjects in the ITT population with genitourinary tract bleeding at baseline and respective post-baseline assessment.
Measure: Number; unit: participants
Arm/Group | IgPro10
Number analyzed (Participants) | 9
participants | 7

5. Secondary Outcome: Regression of Hemorrhage (Nose)
Description: as for outcome 2
Time Frame: 29 days
Population: The number of participants analyzed represents the number of subjects in the ITT population with nose bleeding at baseline and respective post-baseline assessment.
Measure: Number; unit: participants
Arm/Group | IgPro10
Number analyzed (Participants) | 0

6. Secondary Outcome: Regression of Hemorrhage (Internal)
Description: as for outcome 2
Time Frame: 29 days
Population: The number of participants analyzed represents the number of subjects in the ITT population with internal bleeding at baseline and respective post-baseline assessment.
Measure: Number; unit: participants
Arm/Group | IgPro10
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to Platelet Response
Description: Median time to reach a platelet count ≥ 50 x 10^9/L.
Time Frame: 29 days
Population: ITT analysis. The ITT population comprised all subjects who received at least once study medication.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | IgPro10
Number analyzed (Participants) | 57
days | 2.5 [1.0 to 5.0]

8. Secondary Outcome: Duration of Platelet Response
Description: The number of days the platelet count remained ≥ 50 x 10^9/L.
Time Frame: up to 29 days
Population: Analyzed for responders in the ITT population, i.e., only subjects with at least one platelet measurement ≥ 50 x 10^9/L after start of treatment
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: Responders
Arm/Group | IgPro10
Number analyzed (Participants) | 57
Number analyzed (Responders) | 48
days | 15.4 [8.8 to 21.9]

9. Secondary Outcome: Maximum Platelet Level
Description: Maximum absolute platelet count achieved over the duration of the study.
Time Frame: 29 days
Population: ITT analysis. The ITT population comprised all subjects who received at least once study medication.
Measure: Median (Full Range); unit: 10^9/L
Arm/Group | IgPro10
Number analyzed (Participants) | 57
10^9/L | 154 [10 to 1049]

ADVERSE EVENTS:
Time Frame: 28 Days
Arm/Group | IgPro10
Serious Adverse Events (participants affected / at risk) | 3/57
Other Adverse Events (participants affected / at risk) | 52/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro10 (N=57)
Dizziness (Nervous system disorders) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro10 (N=57)
Headache (Nervous system disorders) | 38 (53)
Pyrexia (General disorders) | 14 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (22)
Contusion (Injury, poisoning and procedural complications) | 10 (11)
Petechiae (Skin and subcutaneous tissue disorders) | 7 (9)
Nausea (Gastrointestinal disorders) | 6 (8)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 6 (8)
Vomiting (Gastrointestinal disorders) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Hyperthermia (General disorders) | 5 (7)
Bilirubin conjugated increased (Investigations) | 5 (5)
Blood bilirubin unconjugated increased (Investigations) | 5 (5)
Mouth haemorrhage (Gastrointestinal disorders) | 4 (10)
Coombs direct test positive (Investigations) | 4 (5)
Gingival bleeding (Gastrointestinal disorders) | 4 (5)
Anisocytosis (Blood and lymphatic system disorders) | 3 (5)
Blood lactate dehydrogenase increased (Investigations) | 3 (3)
Coombs test positive (Investigations) | 3 (3)
Haematocrit decreased (Investigations) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must provide a copy of any results communication to the sponsor for review at least 30 days prior to public release. The sponsor may request any changes necessary to prevent forfeiture of patent rights to data not in the public domain. For a multi-center study, the investigator must wait (i) at least 1 year after the study is completed at all sites or (ii) until notified by the sponsor that no multi-center publication is planned before seeking publication review.